CLINICAL TRIAL: NCT00481962
Title: Health Economic Assessment of Tygacil® in the Treatment of Secondary Peritonitis in Intensive Care Units
Brief Title: Health Economic Assessment of Tygacil® in the Treatment of Secondary Peritonitis in Intensive Care Units (ICUs)
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 3074A1-102184
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Peritonitis
MeSH Terms: conditions — Peritonitis | interventions — Tigecycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Tygacil — Initial dose of 100mg followed by 50mg every 12 hours for 5 to 14 days

SUMMARY:
The main goals of the study are: Assessment of Tygacil's cost-effectiveness; Process cost analysis from a hospital perspective (including length of stay, treatment costs, side effect management costs, costs of monitoring, costs of diagnostic procedures, cost of care (TISS 10 score etc.); Efficacy of Tygacil under usual care conditions (cure rate).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of secondary peritonitis
* Treatment in an ICU
* Patient age >18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinical
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com
Locations (1):
- Multiple Cities, Germany